CLINICAL TRIAL: NCT01552629
Title: A Randomized, Double-blind, Placebo Controlled, Parallel Group, Proof of Concept Study Evaluating the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of QGE031 in the Treatment of Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study Evaluating the Safety and Efficacy of QGE031 in Atopic Dermatitis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQGE031X2201; 2011-002112-84 (EudraCT Number)
Record Dates: First submitted 2012-01-26; First posted 2012-03-13 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Atopic eczema; Skin Diseases; QGE031
MeSH Terms: conditions — Dermatitis, Atopic; Skin Diseases | interventions — ligelizumab; Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Group 1 QGE031 (Experimental): QGE031 will be administered as a subcutaneous dose q2 weeks
  Interventions: Drug: QGE031
- Group 2 Placebo (Placebo Comparator): A QGE031 matched placebo will be administered as a subcutaneous dose q2 weeks
  Interventions: Drug: Placebo
- Group 3 Cyclosporine A (Experimental): Cyclosporine A will be administered (as per label) for atopic dermatitis.
  Interventions: Drug: Cyclosporine A

INTERVENTIONS:
Drug: QGE031
  Arms: Group 1 QGE031
Drug: Placebo
  Arms: Group 2 Placebo
Drug: Cyclosporine A
  Arms: Group 3 Cyclosporine A

SUMMARY:
The study will assess the safety and efficacy of QGE031 in the treatment of moderate to severe atopic dermatitis patients. In addition, QGE031 levels in the blood will be measured and the effect of QGE031 on markers in the blood and skin will be evaluated. Comparisons of the effect of QGE31 will be made with placebo and also cyclosporine, a treatment already established as being effective in atopic dermatitis.

ELIGIBILITY:
Key Inclusion criteria:

* Male and female patients 18 to 65 years of age inclusive (at the time of the screening visit), and who passed screening examinations by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests.
* Presence of atopic dermatitis confirmed by itchy skin condition in the past 12 months (must have), plus three, or more, of the following:

  1. History of involvement of the skin creases (fronts of elbows, behind knees, fronts of ankles, around neck or around eyes)
  2. Personal history of asthma or hay fever
  3. History of generally dry skin in the past year
  4. Onset before age of 2 years
  5. Visible flexural dermatitis
* Patients with an EASI score of ≥20 at screening and stable AD (not currently experiencing an acute flare of their AD or had a significant change in the extent of their disease or their treatment regimen in the month prior to enrollment)
* Patients with a Total IgE in the range of 30 to 5000 IU/mL inclusive

Key exclusion criteria:

* Pregnant or nursing (lactating) women, where pregnancy was defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners had been sterilized by vasectomy or other means unless they were using a highly effective method of birth control:
* Total abstinence
* Male/female sterilization
* Combination of any two of the following (a+b or a+c or b+c):

  1. Use of oral, injected or implanted hormonal methods of contraception
  2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-01-05 (Actual); Primary Completion 2013-08-28 (Actual); Study Completion 2013-08-28 (Actual)

PRIMARY OUTCOMES:
Change in Eczema Area and Severity Index(EASI) | baseline, 12 weeks
  Efficacy response will be assessed using EASI.

SECONDARY OUTCOMES:
Change in Investigator Global Assessment (IGA) for atopic dermatitis | 6 weeks, 12 weeks
  Participants dermatitis will be visually assessed and an IGA score will be determined by the Investigator using a prespecified evaluation criteria.
Number of participants with adverse events | 24 weeks
  Adverse events will be determined by observation and non-leading questioning of patients, and by measuring safety parameters (electrocardiograms, clinical laboratory, blood pressure)
QGE031 plasma concentrations | 24 weeks
  Blood samples will be collected on Day 1(predose),15, 29, 43, 57, 71, 85, 99, 113, 127, 141, 155, and 169 for determination of QGE031 serum levels

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Nice, France
- Germany (2):
  - Novartis Investigative Site, Kiel, Germany
  - Novartis Investigative Site, Bonn

REFERENCES:
- See also: Abstract for CQGE031X2201 — http://onlinelibrary.wiley.com/doi/10.1111/exd.13200/epdf